CLINICAL TRIAL: NCT01050088
Title: Effectiveness of Sucrose Analgesia in Infants Undergoing Casting for Club Foot
Brief Title: Sucrose Analgesia in Infants Undergoing Casting for Club Foot
Acronym: SCF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Weigl Daniel MD, Schneider Children's MedicalCenter in Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 005411
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Clubfoot
Keywords: clubfoot; casting; ponseti; discomfort
MeSH Terms: conditions — Clubfoot | interventions — sodium lactobionate sucrose solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose (Experimental): 5cc sucrose solution
  Interventions: Dietary Supplement: sucrose solution
- Saline (Placebo Comparator): 5cc saline p/o
  Interventions: Dietary Supplement: Saline

INTERVENTIONS:
Dietary Supplement: sucrose solution — 5cc 5% sucrose solution P/O
  Arms: Sucrose
Dietary Supplement: Saline — 5cc saline p/o
  Other Names: 5cc Saline solution
  Arms: Saline

SUMMARY:
Babies with congenital clubfeet are treated by the Ponseti casting method. The procedure may cause discomfort to the patient. This study will examine the use of 5 CC Sucrose solution as a comforting agent for the babies.

DETAILED DESCRIPTION:
Babies who were born with congenital clubfeet are currently being treated by the conventional Ponseti method. This procedure is done in an outpatient clinic setup. The procedure is painless but may cause some discomfort to the patient. This study will examine the use of 5 CC Sucrose solution as a comforting agent for the babies. The control group will consist of patients who will get 5cc saline pre cast application, while the study group will be given 5cc of Sucrose solution. Patients and physicians are blinded to the treatment they get. Outcome measures will include pulse rate and oxygenation as an accepted measure of discomfort.

ELIGIBILITY:
Inclusion Criteria:

* All otherwise healthy babies who need casting for congenital clubfeet

Exclusion Criteria:

* All non idiopathic conditions for clubfoot, all individuals who have any kind of known systemic illness, all babies born to diabetic mothers.

Ages: 4 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Pulse rate, Blood oxygenation | During casting

CONTACTS AND LOCATIONS:
Overall Officials: Danielw M Weigl, MD, Principal Investigator — Schneider Children's Medical Center; Kalman Katz, Prof., Study Director — Schneider Children's Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel